CLINICAL TRIAL: NCT06065267
Title: Efficacy of Two-week Therapy With Levofloxacin-based Concomitant Regimen Versus Levofloxacin-based Sequential Regimen for Helicobacter Pylori Infection in Syrian Population: a Prospective Single-center Randomized Controlled Trial
Brief Title: Levofloxacin Concomitant Versus Levofloxacin Sequential
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Damascus Hospital (Other)
Responsible Party: Principal Investigator, Marouf Alhalabi, head of digestive diseases department, Damascus Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G-9-23
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; levofloxacine; concomitant; sequential
MeSH Terms: interventions — Esomeprazole; Ofloxacin; Metronidazole; Amoxicillin; Levofloxacin; Tablets; Omeprazole

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sequential (Experimental): Measure eradication rate of Helicobacter pylori infection with Levofloxacien sequential based regimen
  Interventions: Drug: sequential
- concomitant (Active Comparator): Measure eradication rate of Helicobacter pylori infection with Livofloxacine concomitant based regimen
  Interventions: Drug: Levofloxacin 500Mg Oral Tablet

INTERVENTIONS:
Drug: sequential — amoxicillin 1000 mg bid ,esomprazole 20 bid for one week then levofloxacine 500 mg q.d, metraonidazoel 500 500 bid, and esomprazole 20 bid for one week
  Other Names: Esomeprazole; levofloxacine; metronidazole; amoxicillin
  Arms: sequential
Drug: Levofloxacin 500Mg Oral Tablet — Levofloxacin 500 mg qd, amoxicillin 500 2cab bid,Tinadizole 500 bid, esomprazole 20 bid
  Other Names: Amoxicilline; Esomeprazol; Tinadizole
  Arms: concomitant

SUMMARY:
The goal of this trial is to determine the efficacy of levofloxacin based sequential treatment regimen or concomitant levofloxacin based regimens as empirical first-line therapy in the Syrian population

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged greater than 18 years old who have H. pylori infection diagnosed by any of following three methods:
* Positive rapid urease test (CLOtest).
* Histologic evidence of H. pylori by modified Giemsa staining.
* Positive 13C-urea breath test. without prior eradication therapy and are willing to receive therapy.

Exclusion Criteria:

* Children and teenagers aged less than 18 years.
* Previous eradication treatment for H. pylori.
* Patients who took any drug, which could influence the study results such as proton pump inhibitor, H2 blocker, mucosal protective agent and antibiotics.
* History of gastrectomy.
* Gastric malignancy, including adenocarcinoma and lymphoma,
* Previous allergic reaction to antibiotics (Amoxicillin, Tinadizole,
* Doxycycline,Bismuth subsalicylate,) and prompt pump inhibitors (Es- omeprazole).
* Contraindication to treatment drugs.
* Pregnant or lactating women.
* Severe concurrent disease.
* Liver cirrhosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori infection | 8 week from begning of treatment
  Eradication rate of Helicobacter infected patients

CONTACTS AND LOCATIONS:
Overall Officials: Marouf M Alhalabi, MD, Principal Investigator — general assambly of damascus hospital
Locations (1):
- General Assembly of Damascus Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alhalabi M, Almokdad R. Efficacy of a 2-week therapy with levofloxacin concomitant versus a levofloxacin sequential regimen for Helicobacter pylori infection in the Syrian population: a study protocol for randomized controlled trial. Trials. 2024 Jan 15;25(1):55. doi: 10.1186/s13063-024-07906-3. PMID 38225650